CLINICAL TRIAL: NCT00113620
Title: A Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of Dextromethorphan and Quinidine at Two Dose Levels in the Treatment of the Pain of Diabetic Neuropathy
Brief Title: Safety and Efficacy of Dextromethorphan and Quinidine in the Treatment of the Pain of Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-AVR-109
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Pain; Diabetic Neuropathy
Keywords: distal symmetrical; pain; lower extremities; dextromethorphan
MeSH Terms: conditions — Pain; Diabetic Neuropathies

INTERVENTIONS:
Drug: Neurodex

SUMMARY:
The purpose of this study is to determine whether dextromethorphan (Neurodex) and quinidine are effective in the treatment of pain of diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Established diabetic therapy for at least 3 months
* Lab-supported diagnosis of painful diabetic distal symmetric sensory/motor polyneuropathy
* Pain the previous three months
* Not pregnant

Exclusion Criteria:

* Patient failed adequate trial of 3 or more medications or has required narcotics for pain
* History of torsades de pointes
* Sensitivity to quinidine or opiate drugs (codeine, etc)
* Severe pain that could confound the assessment
* Patient has had any amputations
* Patient has participated in the past 30 days or is currently participating in another trial
* Patient has previously received treatment with dextromethorphan and quinidine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Pain rating scale obtained from patient diaries

SECONDARY OUTCOMES:
Additional diary rating scales and scores obtained from clinic visits

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Pivotal Research Centers, Mesa, Arizona
  - Dedicate Clinical Research, Inc., Sun City, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Research Solutions, Jonesboro, Arkansas
  - Bay Area Foot Care, Castro Valley, California
  - South Bay Clinical Research Inc., Inglewood, California
  - Pacific Sleep Medicine Services, Inc., Los Angeles, California
  - Pacific Sleep Medicine Services, Inc., Palm Springs, California
  - Northern California Research Group, Sacramento, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - University Clinical Research - DeLand, DeLand, Florida
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Laszlo J. Mate, MD, West Palm Beach, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - Investigative Clinical Reserach of Indiana, LLC, Indianapolis, Indiana
  - Crossroads Research, Inc., Owings Mills, Maryland
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Radiant Research - St. Louis, St Louis, Missouri
  - Montana Neuroscience Institute, Missoula, Montana
  - Creighton Diabetes Center, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Upstate Clinical Research, LLC, Albany, New York
  - DiGiovanna Family Care Center, Great Neck, New York
  - Weill Medical College of Cornell University - Peripheral Neuropathy Center, New York, New York
  - Vital Research, Greensboro, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Radiant Research - Akron, Mogadore, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - Knights Road Medical, Bensalem, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research - Greer, Greer, South Carolina
  - Radiant Research, Dallas, Texas
  - Nerve & Muscle Center of Texas, Houston, Texas
  - Diabetes & Glandular Disease Research Assoc., San Antonio, Texas
  - SAM Clinical Research, San Antonio, Texas
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - University of Wisconsin Medical School, Madison, Wisconsin

REFERENCES:
- [Result] Shaibani AI, Pope LE, Thisted R, Hepner A. Efficacy and safety of dextromethorphan/quinidine at two dosage levels for diabetic neuropathic pain: a double-blind, placebo-controlled, multicenter study. Pain Med. 2012 Feb;13(2):243-54. doi: 10.1111/j.1526-4637.2011.01316.x. Epub 2012 Feb 7. PMID 22314263